CLINICAL TRIAL: NCT03203018
Title: Health Literacy and Cardiovascular Knowledge Workshop in Women From Disadvantaged Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Director of Linda Joy Pollin Cardiovascular Wellness Center for Women, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 235HLT-HMO-CTIL
Record Dates: First submitted 2017-06-26; First posted 2017-06-29 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Health Literacy; Communication
Keywords: Cardiovascular Diseases (CVD); Community-based intervention; Socio-economic status (SES); Health literacy (HL)
MeSH Terms: conditions — Communication; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This is a pre/post study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women participating in HL intervention (Experimental): Groups of women from disadvantaged communities will participate in a three session health literacy workshop
  Interventions: Behavioral: Interactive workshop based on community specific needs

INTERVENTIONS:
Behavioral: Interactive workshop based on community specific needs — Intervention components will include lecture on women's CVD, workshop on how to prepare for a doctor's visit, patient's rights and patient-doctor communication skills, and a "know your numbers" workshop, including understanding blood test results.

SUMMARY:
The current health literacy (HL) pilot intervention was designed through focus groups with women in low socio-economic status (SES) communities. The primary HL issue identified was communication challenges at doctors' visits. As a unique HL intervention tailored to the participants' preferences, this intervention can serve as a model for improving HL in similar communities worldwide.

Objectives include increasing the percentage of women who utilize patient-doctor communication skills and increasing their cardiovascular disease (CVD) knowledge. A unique HL intervention tailored to the participants' preferences was designed which consisted of three workshops conducted in municipality-sponsored women's groups in low SES Jerusalem communities. Questionnaires were completed before and three months after the intervention. The study answers the following: Can HL workshops improve patient-doctor communication skills and CVD knowledge in low SES women?

DETAILED DESCRIPTION:
The current health literacy (HL) pilot intervention was designed through focus groups with women in low socio-economic status (SES) communities. The primary HL issue identified was communication challenges at doctors' visits. As a unique HL intervention tailored to the participants' preferences, this intervention can serve as a model for improving HL in similar communities worldwide.

Objectives include increasing the percentage of women who utilize patient-doctor communication skills, prepare for their doctor's visit, and increase their cardiovascular disease (CVD) knowledge.

In order to accomplish these objectives, a unique HL intervention tailored to the participants' preferences was designed which consisted of three workshops conducted in municipality-sponsored women's groups in low SES Jerusalem communities. This intervention consisted of a three consecutive weekly workshop conducted in women's support groups in disadvantaged communities in Jerusalem. The workshop includes women's heart health sessions, as well as sessions about how to make the most of a doctor's visit, which includes role play and teach back method practice. A self-admitted questionnaire regarding CVD and relevant HL knowledge and behaviors was completed at the beginning of the intervention, and three months after the last session.

This study answers the question of whether a three session HL workshop for women can successfully raise their CVD knowledge and awareness, as well as change behaviors of women in terms of preparing for doctor's visits.

ELIGIBILITY:
Inclusion Criteria:

* Women from Jerusalem
* Hebrew and Arabic speakers

Exclusion Criteria:

* None

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in preparation for doctor's visit | Before intervention and three months after intervention
  Women complete self report survey indicating if whether or not they prepared for their doctor's visit, whether or not they prepared a list of questions for their doctor's visit, a list of symptoms, a list of medications, and their medical background information

SECONDARY OUTCOMES:
Change in cardiovascular disease knowledge | At baseline and three month after intervention
  Cardiovascular disease knowledge will be assessed through a self report questionnaire based on the American Heart Association's Cardiovascular disease knowledge survey items
Change in perceived efficacy in patient-physician interaction | At baseline and three month after intervention
  Perceived efficacy in patient-physician interaction (PEPPI) will be assessed via PEPPI self report scale (Maly, Frank, Marshall, Diametteo, Reuben, 1998)
Change in knowledge of health measures | At baseline and three month after intervention
  Knowledge of health measures will be assessed through self report questionnaire
Change in reading blood test results | At baseline and three month after intervention
  Reading blood test results will be assessed through self report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Donna Zwas, MD, MPH, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peerson A, Saunders M. Health literacy revisited: what do we mean and why does it matter? Health Promot Int. 2009 Sep;24(3):285-96. doi: 10.1093/heapro/dap014. Epub 2009 Apr 16. PMID 19372101
- [Background] Safeer RS, Keenan J. Health literacy: the gap between physicians and patients. Am Fam Physician. 2005 Aug 1;72(3):463-8. PMID 16100861
- [Background] Institute of Medicine (US) Committee on Health Literacy; Nielsen-Bohlman L, Panzer AM, Kindig DA, editors. Health Literacy: A Prescription to End Confusion. Washington (DC): National Academies Press (US); 2004. Available from http://www.ncbi.nlm.nih.gov/books/NBK216032/ PMID 25009856
- [Background] Williams MV, Davis T, Parker RM, Weiss BD. The role of health literacy in patient-physician communication. Fam Med. 2002 May;34(5):383-9. PMID 12038721
- [Background] Dewalt DA, Berkman ND, Sheridan S, Lohr KN, Pignone MP. Literacy and health outcomes: a systematic review of the literature. J Gen Intern Med. 2004 Dec;19(12):1228-39. doi: 10.1111/j.1525-1497.2004.40153.x. PMID 15610334
- [Background] Baker DW, Parker RM, Williams MV, Clark WS. Health literacy and the risk of hospital admission. J Gen Intern Med. 1998 Dec;13(12):791-8. doi: 10.1046/j.1525-1497.1998.00242.x. PMID 9844076
- [Background] Martin LR, Williams SL, Haskard KB, Dimatteo MR. The challenge of patient adherence. Ther Clin Risk Manag. 2005 Sep;1(3):189-99. PMID 18360559
- [Derived] Greenberg KL, Leiter E, Donchin M, Agbaria N, Karjawally M, Zwas DR. Cardiovascular health literacy and patient-physician communication intervention in women from disadvantaged communities. Eur J Prev Cardiol. 2019 Nov;26(16):1762-1770. doi: 10.1177/2047487319853900. Epub 2019 Jun 12. PMID 31189377